CLINICAL TRIAL: NCT02348359
Title: A Randomized, Double-Masked, Placebo-Controlled, Dose- Finding, Non-Inferiority Study of X-82 Plus Prn Intravitreal (Ivt) Anti-VEGF Compared to Prn Ivt Anti-VEGF Monotherapy in Neovascular AMD
Brief Title: X-82 to Treat Age-related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis found study had achieved primary objective
Sponsor: Tyrogenex (Industry)
Collaborators: SynteractHCR (Industry); International Drug Development Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X82-OPH-201
Record Dates: First submitted 2015-01-21; First posted 2015-01-28 (Estimated); Results first posted 2018-06-27 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: Age-Related Macular Degeneration (AMD); Macular Degeneration; Exudative Age-related Macular Degeneration; AMD; Macular Degeneration, Age-related, 10; Eye Diseases; Retinal Degeneration; Retinal Diseases
Keywords: Vascular Endothelial Growth Factor (VEGF); Platelet Derived Growth Factor (PDGF); AMD
MeSH Terms: conditions — Macular Degeneration; Macular Degeneration, Age-Related, 10; Eye Diseases; Retinal Degeneration; Retinal Diseases | interventions — aflibercept; Ranibizumab; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 50 mg of X-82 plus ivt anti-VEGF prn (Experimental): Subject will administer one 50 mg tablet of X-82 and one placebo tablet once daily. Subjects will be assessed for the need for retreatment with ivt anti-VEGF therapy at each visit.
  Interventions: Drug: X-82; Drug: Anti-VEGF
- 100 mg of X-82 plus ivt anti-VEGF prn (Experimental): Subject will administer two 50 mg tablets of X-82 once daily. Subjects will be assessed for the need for retreatment with ivt anti-VEGF therapy at each visit.
  Interventions: Drug: X-82; Drug: Anti-VEGF
- 200 mg of X-82 plus ivt anti-VEGF prn (Experimental): Subject will administer two 100 mg tablets of X-82 once daily. Subjects will be assessed for the need for retreatment with ivt anti-VEGF therapy at each visit.
  Interventions: Drug: X-82; Drug: Anti-VEGF
- Placebo plus ivt anti-VEGF prn (Placebo Comparator): Subject will administer two placebo tablets once daily. Subjects will be assessed for the need for retreatment with ivt anti-VEGF therapy at each visit.
  Interventions: Drug: Anti-VEGF; Drug: Placebo

INTERVENTIONS:
Drug: X-82
  Other Names: X-82 tablets
  Arms: 100 mg of X-82 plus ivt anti-VEGF prn; 200 mg of X-82 plus ivt anti-VEGF prn; 50 mg of X-82 plus ivt anti-VEGF prn
Drug: Anti-VEGF
  Other Names: Aflibercept (Eylea); Ranibizumab (Lucentis); Bevacizumab (Avastin)
Drug: Placebo
  Arms: Placebo plus ivt anti-VEGF prn

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of X-82 in the treatment of vision loss due to wet AMD.

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1:1:1 ratio to the following dose groups:

* X-82 50 mg plus ivt anti-VEGF prn
* X-82 100 mg plus ivt anti-VEGF prn
* X-82 200 mg plus ivt anti-VEGF prn
* Placebo plus ivt anti-VEGF prn

Subjects will be treated for a total of 52 weeks with one of three doses of X-82 or placebo.

Primary Efficacy Outcome:

The primary efficacy outcome is the change in visual acuity score from Day -1 to 52 Weeks after randomization.

Safety Outcomes:

Systemic and ocular safety will be evaluate by assessing ECG, laboratory analyses, adverse events and serious adverse events.

Approximately 132 subjects will be randomized into one of the four arms (33 subjects per dose group).

ELIGIBILITY:
Inclusion Criteria:

* Participants mush have wet AMD which has been diagnosed and treated with anti-VEGF in one or both eyes for at least 6 months prior to joining the study and has required at least two prior injections of intravitreal (ivt) anti-VEGF at intervals of not greater than 6 weeks for the past two injections in the eye that is selected to be the study eye.
* Must have demonstrated a reduction in macular fluid or macular thickness in the study eye 14 days following an anti-VEGF injection at Screening Visit 1
* Early Treatment Diabetic Retinopathy (ETDRS) Best Corrected Visual Acuity (BCVA) of 25 letters (20/320) or better in both eyes

Exclusion Criteria:

* Previous vitrectomy to the study eye within 30 days of Screening Visit 1
* Choroidal neovascularization (CNV) due to causes other than AMD
* Proliferative diabetic retinopathy in either eye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-03-16 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel E Salazar, PhD, Principal Investigator — Study PI
Locations (35):
- United States (35):
  - Tucson, Arizona
  - Beverly Hills, California
  - Huntington Beach, California
  - Redlands, California
  - Sacramento, California
  - Colorado Springs, Colorado
  - Golden, Colorado
  - New London, Connecticut
  - Fort Myers, Florida
  - Lakeland, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Palm Beach Gardens, Florida
  - Augusta, Georgia
  - Lemont, Illinois
  - Oak Forest, Illinois
  - Indianapolis, Indiana
  - Baltimore, Maryland
  - Glen Burnie, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Portsmouth, New Hampshire
  - Bloomfield, New Jersey
  - Albany, New York
  - New York, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Youngstown, Ohio
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Houston, Texas
  - The Woodlands, Texas
  - Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 39 sites in the United States. There were 36 sites that screened subjects and 3 sites that did not screen any subjects. A total of 157 subjects were randomly assigned and treated in the study.
Groups:
- 50 mg of X-82 Plus Ivt Anti-VEGF Prn: Subject will administer one 50 mg tablet of X-82 and one placebo tablet once daily. Subjects will be assessed for the need for retreatment with ivt anti-VEGF therapy at each visit.
  X-82
  Anti-VEGF
- 100 mg of X-82 Plus Ivt Anti-VEGF Prn: Subject will administer two 50 mg tablets of X-82 once daily. Subjects will be assessed for the need for retreatment with ivt anti-VEGF therapy at each visit.
  X-82
  Anti-VEGF
- 200 mg of X-82 Plus Ivt Anti-VEGF Prn: Subject will administer two 100 mg tablets of X-82 once daily. Subjects will be assessed for the need for retreatment with ivt anti-VEGF therapy at each visit.
  X-82
  Anti-VEGF
- Placebo Plus Ivt Anti-VEGF Prn: Subject will administer two placebo tablets once daily. Subjects will be assessed for the need for retreatment with ivt anti-VEGF therapy at each visit.
  Anti-VEGF
  Placebo
Period: Overall Study
Arm/Group | 50 mg of X-82 Plus Ivt Anti-VEGF Prn | 100 mg of X-82 Plus Ivt Anti-VEGF Prn | 200 mg of X-82 Plus Ivt Anti-VEGF Prn | Placebo Plus Ivt Anti-VEGF Prn
Started | 40 | 39 | 39 | 39
Completed | 29 | 22 | 25 | 27
Not Completed | 11 | 17 | 14 | 12

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | 50 mg of X-82 Plus Ivt Anti-VEGF Prn | 100 mg of X-82 Plus Ivt Anti-VEGF Prn | 200 mg of X-82 Plus Ivt Anti-VEGF Prn | Placebo Plus Ivt Anti-VEGF Prn | Total
Number analyzed (Participants) | 40 | 39 | 39 | 39 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (8.23) | 73.5 (8.33) | 75.0 (7.63) | 75.9 (7.65) | 75.0 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 16 | 18 | 23 | 79
  Male | 18 | 23 | 21 | 16 | 78
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 40 | 38 | 38 | 38 | 154
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 39 | 39 | 39 | 157
Best corrected visual acuity [Mean (Standard Deviation); unit: Number of letters] | 72.3 (9.41) | 71.2 (12.17) | 71.9 (13.17) | 68.8 (12.43) | 71.0 (11.83)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity Score From Day -1 to Week52
Description: The primary outcome is the change in the visual acuity score from Day -1 to 52 weeks after randomization.
Time Frame: Week 52
Population: Analysis restricted to subjects who completed 52 weeks of treatment
Measure: Mean (Standard Deviation); unit: number of letters
Arm/Group | 50 mg of X-82 Plus Ivt Anti-VEGF Prn | 100 mg of X-82 Plus Ivt Anti-VEGF Prn | 200 mg of X-82 Plus Ivt Anti-VEGF Prn | Placebo Plus Ivt Anti-VEGF Prn
Number analyzed (Participants) | 23 | 19 | 17 | 22
number of letters | 0.2 (4.14) | -0.9 (6.57) | 1.7 (5.58) | -0.3 (10.63)

ADVERSE EVENTS:
Time Frame: All adverse events were collected and reported from time of participant study entry until discharge of last participant from the study. Individual subject participation in the study ranged from 0-14 months
Arm/Group | 50 mg of X-82 Plus Ivt Anti-VEGF Prn | 100 mg of X-82 Plus Ivt Anti-VEGF Prn | 200 mg of X-82 Plus Ivt Anti-VEGF Prn | Placebo Plus Ivt Anti-VEGF Prn
All-Cause Mortality (participants affected / at risk) | 0/40 | 1/39 | 0/39 | 0/39
Serious Adverse Events (participants affected / at risk) | 6/40 | 7/39 | 3/39 | 2/39
Other Adverse Events (participants affected / at risk) | 39/40 | 38/39 | 37/39 | 34/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 50 mg of X-82 Plus Ivt Anti-VEGF Prn (N=40) | 100 mg of X-82 Plus Ivt Anti-VEGF Prn (N=39) | 200 mg of X-82 Plus Ivt Anti-VEGF Prn (N=39) | Placebo Plus Ivt Anti-VEGF Prn (N=39)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
sudden cardiac death (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endopthalmitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
B cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 50 mg of X-82 Plus Ivt Anti-VEGF Prn (N=40) | 100 mg of X-82 Plus Ivt Anti-VEGF Prn (N=39) | 200 mg of X-82 Plus Ivt Anti-VEGF Prn (N=39) | Placebo Plus Ivt Anti-VEGF Prn (N=39)
Atrioventricular block (Cardiac disorders) | 3 | 1 | 2 | 3
Supraventricular systole (Cardiac disorders) | 2 | 2 | 0 | 0
Conjunctival hemorrhage (Eye disorders) | 2 | 2 | 2 | 2
Vitreous detachment (Eye disorders) | 3 | 2 | 2 | 1
Cataract (Eye disorders) | 2 | 1 | 2 | 2
Retinal hemorrhage (Eye disorders) | 2 | 2 | 1 | 1
Dry eye (Eye disorders) | 0 | 1 | 2 | 2
Visual acuity reduced (Eye disorders) | 2 | 2 | 1 | 0
Neovascular age related macular degeneration (Eye disorders) | 1 | 0 | 0 | 3
Vitreous floaters (Eye disorders) | 2 | 2 | 0 | 0
Diplopia (Eye disorders) | 2 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0 | 2
Photopsia (Eye disorders) | 0 | 2 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 2 | 0
Eye pain (Eye disorders) | 0 | 2 | 0 | 0
Eyelash discoloration (Eye disorders) | 0 | 0 | 2 | 0
Metamorphopsia (Eye disorders) | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 9 | 2
nausea (Gastrointestinal disorders) | 6 | 2 | 1 | 1
vomiting (Gastrointestinal disorders) | 3 | 2 | 2 | 1
dyspepsia (Gastrointestinal disorders) | 1 | 2 | 3 | 1
abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 3 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Fatigue (General disorders) | 2 | 4 | 6 | 0
Oedema peripheral (General disorders) | 1 | 1 | 3 | 1
Chest pain (General disorders) | 0 | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 7 | 2 | 5 | 2
Urinary tract infection (Infections and infestations) | 2 | 5 | 1 | 2
Bronchitis (Infections and infestations) | 2 | 2 | 3 | 0
Influenza (Infections and infestations) | 1 | 1 | 3 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2
Diverticulitis (Infections and infestations) | 0 | 2 | 0 | 0
Tinea cruris (Infections and infestations) | 2 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 8 | 11 | 9 | 2
Aspartate aminotransferase increased (Investigations) | 6 | 10 | 8 | 1
Blood pressure increased (Investigations) | 2 | 2 | 4 | 3
Bllod creatinine phosphokinase increased (Investigations) | 1 | 3 | 3 | 2
Blood glucose increased (Investigations) | 2 | 2 | 2 | 1
Hepatic enzyme increase (Investigations) | 1 | 3 | 3 | 0
Platelet count decreased (Investigations) | 1 | 2 | 3 | 1
Urine protein/creatinine ratio increased (Investigations) | 2 | 3 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 3 | 1 | 1
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 2
Weight decreased (Investigations) | 0 | 0 | 3 | 0
White blood cells urine positive (Investigations) | 0 | 1 | 0 | 2
Prostate specific antigen increased (Investigations) | 0 | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 4 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 3 | 5 | 10 | 0
Headache (Nervous system disorders) | 3 | 2 | 4 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 1 | 1
Ageusia (Nervous system disorders) | 0 | 0 | 3 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Hair color change (Skin and subcutaneous tissue disorders) | 2 | 10 | 13 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2 | 6 | 0
Hypertension (Vascular disorders) | 2 | 4 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/59/NCT02348359/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-11): https://cdn.clinicaltrials.gov/large-docs/59/NCT02348359/SAP_001.pdf